CLINICAL TRIAL: NCT01419977
Title: Randomized Double Blind Placebo Controlled Treatment of Sickle Cell Patients Hospitalized in Pain Crisis With Prophylactic Dose LMWH Versus Placebo
Brief Title: Treatment of Sickle Cell Patients Hospitalized in Pain Crisis With Prophylactic Dose Low-molecular-weight Heparin (LMWH) Versus Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eisai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00023305
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: sickle cell disease; vaso-occlusive crisis; anticoagulation
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Normal saline solution
  Interventions: Drug: Placebo
- Dalteparin (Experimental): 5000 unites subcutaneously, Other Name: Fragmin
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Placebo — Normal saline solution, administered by nursing staff once daily
  Arms: Placebo
Drug: Dalteparin — Low molecular weight heparin (LMWH), 5000 unites subcutaneously, administered by nursing staff once daily, Other Name: Fragmin
  Arms: Dalteparin

SUMMARY:
Sickle cell disease (SCD) is one of the most common inherited diseases worldwide and exhibits highest frequency in people of African descent. Patients with SCD currently have few treatment options, with hydroxyurea being the only medication approved to reduce the frequency of vaso-occlusive crisis (VOC) and prevent other SCD complications such as acute chest syndrome. Once patients develop VOC, hospitalizations aim to alleviate pain; no specific therapy is currently available to otherwise affect the course of the VOC. However, there has been increasing interest in the role of coagulation in the pathogenesis of SCD. The investigators hypothesize that low dose anticoagulant therapy, such as prophylactic dose low-molecular-weight heparin (LMWH), could be a novel way to ameliorate the vaso-occlusive process and thereby hasten the resolution of pain.

DETAILED DESCRIPTION:
This is a double blind prospective randomized placebo controlled study with an enrollment target of 100 patients. All subjects with SCD that meet inclusion criteria while inpatient, will be eligible for the study and randomized to receive prophylactic LMWH or placebo. Treatment with either LMWH (dalteparin 5000 IU subcutaneously daily) or placebo will occur for the initial 7 days of hospitalization. Randomization will occur within Investigational Drug Services, which will dispense and label medications to all patients. All patients will be followed throughout their hospitalization as well as in the outpatient clinic. The initial blood sample will be obtained within 36 hours of admission.

Following randomization, blood will be drawn to perform: D-dimer, prothrombin fragment 1.2, thrombin-antithrombin complex, and Thrombin Generation Assay (TGA). Blood will be drawn as an inpatient (at admission, day 3, and day 5), as well as during a single outpatient follow-up visit two weeks post discharge. Patients with prolonged hospitalization will only have blood drawn on admission, day 3, and day 5, with a final blood draw as an outpatient (at least 14 days after discharge). Treatment by prophylactic LMWH or placebo will occur for the initial 7 days of hospitalization or until discharge.

Clinical pain scores will be performed twice daily throughout for the initial 7 days of hospitalization of all patients. The primary pain assessment tool will be a 10-cm horizontal visual analog scale (VAS), with "0" corresponding to no pain at one end and "10" indicating the worst pain at the other. The VAS test will be administered by the same blinded study coordinator or PI throughout the study, using standardized instructions. Pain will also be assessed during the follow up outpatient visit (to confirm patient's pain has returned to their baseline).

Patients will be recommended to follow up in outpatient clinic approximately 2-4 week following hospitalization. At this time, patients will be examined, have their clinical pain score determined, and have final blood draw for testing as detailed above. Should patients not return within 4 weeks, patient will be contacted by phone to determine their clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Documented HgbSS or HgbS-beta0 thalassemia by previous hemoglobin electrophoresis,
* age greater than 18 years old, and
* admit diagnosis of vaso-occlusive crisis.

Labs must be drawn within 36 hours of admission and randomization to treatment arm must occur during this time.

Exclusion Criteria:

* End stage renal disease (creatinine >3.0 mg/dL),
* use of antiplatelet or anticoagulation medication for an alternative indication,
* use of steroids or immunosuppressive medications,
* platelet count less than 100 X 109/L,
* history or development of heparin induced thrombocytopenia, packed red blood cell transfusion in the past one month, or
* recent hospitalization with discharge within the past 1 week.

Patients with re-admissions will not be enrolled again and will have no further samples drawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirmish Shah, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 34 subjects were consented, 29 are received drug and had the day 1 blood draw. 2 subjects withdrew prior to receiving study drug. In addition, 2 subjects were discharged and 1 subject received a transfusion prior to the blood draw on day 1.
Groups:
- Dalteparin: Dalteparin: Low molecular weight heparin (LMWH), 5000 units subcutaneously, administered by nursing staff once daily, Other Name: Fragmin
Period: Overall Study
Arm/Group | Placebo | Dalteparin
Started | 16 | 13
Completed | 16 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dalteparin | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 12 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in D-dimer
Description: Patients will have D-dimer,for samples drawn on Day 1 and Day 3
Time Frame: Day 1 and Day 3
Population: 9 subjects were discharged prior to day 3 so the day 3 blood sample was not obtained.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 11 | 9
ng/mL | 478.8 (312.4) | 260.1 (200.3)

2. Primary Outcome: Change in Clinical Pain Scores
Description: The primary pain assessment tool will be a 10-cm horizontal visual analog scale (VAS), with "0" corresponding to no pain at one end and "10" indicating the worst pain at the other.
Time Frame: Baseline to day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 16 | 13
units on a scale | -0.3 (0.5) | -1.6 (0.4)

3. Primary Outcome: Change in Thrombin Generation Assay - Endogenous Thrombin Potential
Description: Patients will have thrombin generation assay samples drawn on Day 1 and 3
Time Frame: Day 1 and Day 3
Population: 9 subjects were discharged prior to day 3 so the day 3 blood sample was not obtained.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 11 | 9
nM | 13.4 (34.5) | -45.98 (47.31)

4. Primary Outcome: Change in Clinical Pain Scores
Description: as for outcome 2
Time Frame: Baseline to day 3
Population: 9 subjects were discharged prior to obtaining day 3 VAS score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 11 | 9
units on a scale | -0.9 (0.2) | -2.4 (0.9)

ADVERSE EVENTS:
Arm/Group | Placebo | Dalteparin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 0/16 | 0/13

LIMITATIONS AND CAVEATS:
Limitations to our pilot study include the small study sample size, which leads to difficulty in determining significant differences in the outcome measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes